CLINICAL TRIAL: NCT01614431
Title: N Acetyl Cysteine Can Decrease the Progression of Renal Disease in Cystinosis Patients
Brief Title: N Acetyl Cysteine for Cystinosis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Maria Helena Vaisbich, Clinical Professor, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Cystinosis and NAC
Record Dates: First submitted 2012-05-19; First posted 2012-06-08 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2012-06

CONDITIONS: Renal Disease; Cystinosis
Keywords: renal function; before and after N acetyl cysteine; Cystinosis patients
MeSH Terms: conditions — Kidney Diseases; Cystinosis | interventions — Acetylcysteine

ARMS (1):
- N acetyl cysteine (Experimental): NAC will be given to cystinosis patients and we will observe the renal function status and a marker of oxidative stress (TBARS)
  Interventions: Drug: N acetyl cysteine

INTERVENTIONS:
Drug: N acetyl cysteine — N acetyl cysteine to cystinosis patients with CKD stages 1 to 4
  Other Names: N acety cysteine
Drug: N acetyl cysteine — N acetyl cysteine for cystinosis patients CKD stages 1 to 4

SUMMARY:
This study intends to verify the interference of N acetyl cysteine in the progression of chronic kidney disease in patients with Nephropathic Cystinosis.

DETAILED DESCRIPTION:
Patients with Nephropathic Cystinosis have an increased oxidative stress and go to end-stage renal disease, even when all steps of the treatment are done. Therefore, this study is conducted to verify the interference of the stress oxidative in the progression of the renal disease with the use of an oxidant drug, N acetyl cysteine (NAC). The investigators selected patients with good compliance of the treatment. In these patients the investigators evaluate the serum creatinine, creatinine clearance estimated by Schwartz Formula, cystatin C and a marker of oxidative stress, TBARS ( thiobarbituric acid substances). The variables are analyzed 6 months before the introduction of NAC and the three months after NAC.

ELIGIBILITY:
Inclusion Criteria:

* cystinosis patients age under 18 years with good compliance to the treatment with Chronic Kidney Disease 1 to 4 according to KDOQI

Exclusion Criteria:

* patients with CKD stage 5

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2011-03; Primary Completion 2012-01 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
creatinine clearance | change in creatinine clearance evaluated 6 months before , at baseline and after 3 months with NAC
  creatinine clearance will be evaluate 6 months beforw and at baseline and after 3 months with NAC
cystatin c | change in cystatin C from baseline and after 3 months with NAC
  Cystinosis patients will be evaluated 6 months before and at baseline and after 3 months after the use of NAC

CONTACTS AND LOCATIONS:
Overall Officials: Maria Helena Vaisbich, Doctor, Principal Investigator — University of Sao Paulo